CLINICAL TRIAL: NCT02441699
Title: Assessing the Health Impact of a Combined Water and Sanitation Intervention in Rural Odisha, India
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Emory University (Other); KIIT University, Bhubaneswar, Orissa (Unknown); Gram Vikas, Bhubanesar, Orissa (Unknown); Loyola Hospital, Bhubaneswar, Orissa (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 9071
Record Dates: First submitted 2015-04-27; First posted 2015-05-12 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Diarrhea; Enteric Infection; Soil-transmitted Helminth Infection; Stunting
MeSH Terms: conditions — Diarrhea; Growth Disorders | interventions — Sanitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples will be collected and divided into two aliquots. One aliquot will be fixed and used for assessing the rate and intensity of soil-transmitted helminth (STH) infection and the second aliquot will be frozen and used to assess biomarkers of environmental enteropathy and enteric infection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention group: Rural villages in which Gram Vikas has fully implemented its water supply and sanitation (Mantra) intervention. Intervention villages must: 1) be within 3 hours travel to the study office in Brahmapur, 2) have started the intervention by January 2003, and 3) have completed the intervention by January 2013.
  Interventions: Behavioral: Improved water supply and sanitation
- Control group: Rural villages that have been matched with intervention villages on demographics and other criteria. The sampling frame for control villages is limited to those: 1) within 3 hours travel to the study office in Brahmapur, and 2) within Gram Panchayats which do not include an intervention village and are not adjacent to an intervention village, to minimize spillover effects. In addition, both intervention and control villages must appear in the Government of India Census in 2001.

INTERVENTIONS:
Behavioral: Improved water supply and sanitation — Village-level reticulated water supply with distribution to household taps; pour-flush pit latrines.
  Groups: Intervention group

SUMMARY:
This is a matched-cohort study designed to assess the health impact of a rural demand-driven water and sanitation intervention that provides piped treated water and household level pour-flush latrines and bathing rooms, as implemented by Gram Vikas.

DETAILED DESCRIPTION:
We will undertake a matched-cohort study among 84 villages in Ganjam district, Orissa, India to assess the health impact of a program that provides improved water supplies and sanitation to rural villages.

ELIGIBILITY:
Inclusion Criteria:

* Households in participating villages will be eligible to participate in the study if they have at least one child under 5 years.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rural householders living in Ganjam district, Orissa, India.
Sampling Method: Probability Sample
Enrollment: 2940 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Reported diarrhoea in children <5 years | 7-day recall, assessed 4 times during 3-month follow-up rounds

SECONDARY OUTCOMES:
Reported lower respiratory infection in children <5 | 7-day recall, assessed 4 times during 3-month follow-up rounds
Diarrhoea among all ages | 7-day recall, assessed 4 times during 3-month follow-up roundsits
Lower respiratory infection among all ages | 7-day recall, assessed 4 times during 3-month follow-up roundsts
Soil-transmitted helminth infection | Point prevalence assessed in rounds 2 (approximately 90-120 days after study commencement) and 4 (approximately 240 to 360 days after study commencement)
  Stool samples taken and assayed for ascaris, trichuris, hookworm
Height-for-age among children < 2 years | Assessed approximately every 90 days for a total of four measurement over study period
  Children height measured and HAZ scores computed
Weight-for-age among children <5 | Assessed approximately every 90 days for a total of four measurement over study periodAssessed during all four follow up rounds
  Children weighed and WAZ scores computed
Biomarkers of environmental enteropathy and enteric infection | Assessed once during round 3 (approximately 180 to 240 days following commencement of study

CONTACTS AND LOCATIONS:
Locations (1):
- London School of Hygiene & Tropical Medicine, London, United Kingdom

REFERENCES:
- [Derived] Sinharoy SS, Reese HE, Praharaj I, Chang HH, Clasen T. Effects of a combined water and sanitation intervention on biomarkers of child environmental enteric dysfunction and associations with height-for-age z-score: A matched cohort study in rural Odisha, India. PLoS Negl Trop Dis. 2021 Mar 8;15(3):e0009198. doi: 10.1371/journal.pntd.0009198. eCollection 2021 Mar. PMID 33684111
- [Derived] Reese H, Routray P, Torondel B, Sinharoy SS, Mishra S, Freeman MC, Chang HH, Clasen T. Assessing longer-term effectiveness of a combined household-level piped water and sanitation intervention on child diarrhoea, acute respiratory infection, soil-transmitted helminth infection and nutritional status: a matched cohort study in rural Odisha, India. Int J Epidemiol. 2019 Dec 1;48(6):1757-1767. doi: 10.1093/ije/dyz157. PMID 31363748
- [Derived] Reese H, Routray P, Torondel B, Sclar G, Delea MG, Sinharoy SS, Zambrano L, Caruso B, Mishra SR, Chang HH, Clasen T. Design and rationale of a matched cohort study to assess the effectiveness of a combined household-level piped water and sanitation intervention in rural Odisha, India. BMJ Open. 2017 Mar 31;7(3):e012719. doi: 10.1136/bmjopen-2016-012719. PMID 28363920